CLINICAL TRIAL: NCT01202487
Title: Pretreatment of Lacerations With Topical LET (Lidocaine-Epinephrine-Tetracaine) Reduces Pain During Tissue Adhesive Repair in Children: Double-blind, Randomized, Controlled Trial of Efficacy
Brief Title: Gluing Lacerations Utilizing Epinephrine
Acronym: GLUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Stuart Harman, Dr. Stuart Harman MD FRCPC, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6138378804
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Lacerations
Keywords: Laceration; Lacerations; LET; Lidocaine Epinephrine Tetracaine; LAT; Lidocaine Adrenaline Tetracaine; Tissue Adhesive; Skin Glue; Pre-Treatment with LET; Pre-Treatment with LAT; Pre-Treatment with Lidocaine Epinephrine Tetracaine; Pre-Treatment with Lidocaine Adrenaline Tetracaine; Use of LET with Skin Glue; Use of LET with Tissue Adhesive; Histoacryl
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-treatment with LET (Experimental): Pre-treatment with Lidocaine Epinephrine Tetracaine solution at least 45 minutes prior to laceration repair with tissue adhesive
  Interventions: Drug: LET - Lidocaine Epinephrine Tetracaine
- Pre-treatment with Placebo (Placebo Comparator): Pre-treatment with Placebo solution at least 45 minutes prior to laceration repair with tissue adhesive
  Interventions: Drug: LET - Lidocaine Epinephrine Tetracaine

INTERVENTIONS:
Drug: LET - Lidocaine Epinephrine Tetracaine — One time application of 3 cc of Lidocaine Epinephrine Tetracaine Solution at least 45 minutes prior to laceration repair
  Other Names: LAT; Lidocaine Adrenaline Tetracaine

SUMMARY:
Minor lacerations are a commonly treated injury in the paediatric emergency department . Over the past decade, standard closure of these lacerations has evolved from suture repair to closure with tissue adhesive (also referred to as "skin glue"). Local anaesthetic is not routinely used during application of skin glue as it was with sutures. There are, however, several potential advantages to pre-treating wounds with topical LET (Lidocaine-Epinephrine-Tetracaine), a liquid gel with anaesthetic and vasoconstrictive properties. Some believe LET can improve patient comfort, increase the ease of glue application, and lead to better healing when used on lacerations being repaired with tissue adhesive. This study aims to address the question of whether or not pre-treatment with LET improves outcomes in minor lacerations repaired with skin glue. The primary hypothesis is that pre-treatment of minor lacerations with LET will decrease pain (as measured on a Visual Analog Scale) during repair with tissue adhesive.

ELIGIBILITY:
Inclusion Criteria:

* aged 0 to 17 years inclusive;
* with a laceration that is less than 3 cm in length (the upper limit recommended for tissue adhesive repair by the manufacturer).
* with said laceration on the face, torso, trunk or extremities;
* with said laceration deemed by the treating physician to be appropriate for repair via tissue adhesive

Exclusion Criteria:

* the wound for study needs debridement or suturing prior to first glue attempt
* said wound is an animal or human bite or scratch wound, puncture wound, stellate crush wound, wound crossing mucocutaneous junctions, a scalp laceration, an ear laceration, a wound crossing a joint line, a wound on the fingers or toes, or a wound in an area of concentrated hair such as the eyebrow
* the patient has a history of keloid formation or
* a known allergy to cyanoacrylates or
* is presently taking oral steroids, immunostimulants, anticoagulants or other medications known to impair wound healing or haemostasis; or
* has a known diagnosis of Diabetes Mellitus or Vascular Insufficiency

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Pain of Procedure Rating | 2 minutes post-procedure
  Patients will rate the pain experienced during their procedure on a 100 mm Visual Analog Scale (in paitents age 6 and under, parents will rate what pain they believe their child experienced).

SECONDARY OUTCOMES:
Wound Cosmesis | measured at 3 month f/u visit
  Patients will return 3 months post laceration repair for a photograph on their wound. Plastic surgeons blinded to the treatment arm will rate the wound cosmesis via the photographs on a validated 100 mm Visual Analog Scale
Ease of procedure as measured by treating physician | 5 minutes post-procedure
  Immediately after the procedure, the treating physician will rate how easy the repair was on a 100 mm Visual Analog Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart GS Harman, MD FRCPC, Principal Investigator — Children's Hospital of Eastern Ontario; Roger Zemek, MD FRCPC, Study Director — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada